CLINICAL TRIAL: NCT00445003
Title: Intravitreal Ranibizumab or Triamcinolone Acetonide as Adjunctive Treatment to Panretinal Photocoagulation for Proliferative Diabetic Retinopathy
Brief Title: Laser-Ranibizumab-Triamcinolone for Proliferative Diabetic Retinopathy
Acronym: LRTforDME+PRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Genentech, Inc. (Industry); Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-134; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Proliferative Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Diabetic Retinopathy; Diabetic Macular Edema; Lucentis; Ranibizumab; Triamcinolone; Panretinal Photocoagulation; Combination Therapy; pdr
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab; Triamcinolone Acetonide; Adrenal Cortex Hormones; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham injection plus laser (Experimental): Sham injection at baseline and 4 weeks. Focal/grid laser for diabetic macular edema was performed 3 days to 10 days after the injection for all treatment groups.
  Interventions: Behavioral: Sham injection; Procedure: Focal/grid laser
- 0.5mg Ranibizumab plus laser (Experimental): Intravitreal injections of 0.5mg Ranibizumab at baseline and at 4 weeks. Focal/grid laser for diabetic macular edema was performed 3 days to 10 days after the injection for all treatment groups.
  Interventions: Drug: Ranibizumab; Procedure: Focal/grid laser
- 4-mg Triamcinolone Acetonide plus Laser (Active Comparator): 4-mg Triamcinolone Acetonide at baseline and sham injection at 4 weeks. Focal/grid laser for diabetic macular edema was performed 3 days to 10 days after the injection for all treatment groups.
  Interventions: Drug: Triamcinolone Acetonide; Procedure: Focal/grid laser

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of 0.5 mg ranibizumab at baseline and 4 weeks
  Other Names: Lucentis™
  Arms: 0.5mg Ranibizumab plus laser
Drug: Triamcinolone Acetonide — Intravitreal injection of 4 mg triamcinolone acetonide at baseline and sham injection at 4 weeks
  Other Names: corticosteroid
  Arms: 4-mg Triamcinolone Acetonide plus Laser
Behavioral: Sham injection — Sham injection at baseline and 4 weeks
  Arms: Sham injection plus laser
Procedure: Focal/grid laser — Focal/grid laser for diabetic macular edema was performed 3 days to 10 days after the injection for all treatment groups.

SUMMARY:
The purpose of the study is to find out if treatment with an intravitreal injection of triamcinolone or an intravitreal injection of ranibizumab can prevent loss of vision caused by panretinal photocoagulation treatment. At the present time, it is not known whether intravitreal steroid or anti-vascular endothelial growth factor (anti-VEGF) injections are beneficial in preventing vision loss after panretinal photocoagulation (PRP) treatment. It is possible that one or both of the types of injections will prevent vision loss after PRP treatment. However, it is not known whether the benefits of the injections will outweigh the risks. It is possible that because of side effects, the injections may not be as good as laser alone in treating the diabetic retinopathy.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is manifested in retinal neovascularization at the disc (NVD) or elsewhere (NVE). Vitreous hemorrhage or tractional detachment from PDR is a leading cause of severe visual loss and new onset blindness. Without intervention, 60 percent of individuals with diabetic retinopathy will eventually develop PDR, resulting in significant visual loss in nearly fifty percent.

Proliferative diabetic retinopathy is currently treated with panretinal photocoagulation (PRP) which destroys areas of the retina but preserves central vision. PRP is most effectively seen in a regression of new vessels, stabilization of the neovascularization, and reduced risk of visual loss. However, the treatment is associated with unavoidable side effects including macular edema with transient or permanent central vision loss, diminished vision loss, and night vision loss. The treatment applies laser burns to the peripheral retinal tissue, destroying outer photoreceptors and retinal pigment epithelium of the retina, and is thought to exert its effect by increasing oxygen delivery to the inner retina and decreasing viable hypoxic cells which are producing growth factors such as VEGF. Studies have implicated vascular endothelial growth factor (VEGF) as the substance leading to neovascularization and/or increased vascular permeability. Thus, it is reasonable to expect that inhibition of VEGF could reduce both PDR and transient vision loss from macular edema. There are several anti-VEGF drugs. Ranibizumab is the drug to be evaluated in this trial. In one trial of ranibizumab on DME, ten patients with chronic DME received a series of 0.5 mg intraocular injections. The treatments were well tolerated with no ocular or systemic adverse events. Since intraocular injections of ranibizumab significantly reduced foveal thickness and improved visual acuity in all ten patients, there is strong rationale to consider this drug as adjunctive therapy to PRP in a attempt to reduce the acute, transient edema that may occur with PRP.

Similarly, corticosteroids, a class of substances with anti-inflammatory properties, have demonstrated to inhibit the expression of VEGF. Triamcinolone acetonide is often used as a periocular injection for the treatment of cystoid macular edema (CME) secondary to uveitis. Clinically, triamcinolone acetonide is used in the treatment of proliferative vitreoretinopathy and choroidal neovascularization. Studies on patients with proliferative diabetic retinopathy randomly assigned to receive 4 mg triamcinolone 10 to 15 days prior to PRP treatment showed a reduction in central macular thickening, and fluorescein leakage was greater in the injection group than in the control group at 9 and 12 months follow up. Mean visual acuity improved by one line in the injection group and worsened by two lines in the control group.

In summary, there is strong rationale that using either intravitreal ranibizumab or intravitreal triamcinolone acetonide as an adjunct to PRP could reduce the magnitude of vision loss.

This study is being conducted to determine whether intravitreal injection of an anti-VEGF drug or an intravitreal injection of a corticosteroid can reduce the occurrence of macular edema and visual acuity impairment following PRP. Subjects will be randomly assigned with equal probability to one of the following three injection groups:

* Intravitreal injection of 0.5 mg ranibizumab (Lucentis™) at baseline and 4 weeks
* Intravitreal injection of 4 mg triamcinolone acetonide at baseline and sham injection at 4 weeks
* Sham injection at baseline and 4 weeks

The initial injection (or sham) is given on the day of randomization. Focal (macular) photocoagulation is given 7 to 10 days following the injection. Panretinal (scatter) photocoagulation can be initiated either on the same day as the focal photocoagulation (immediately following the focal photocoagulation) or on a subsequent day but must be initiated within 14 days of the baseline injection. Required follow-up visits occur at 4, 14, 34 and 56 weeks.

ELIGIBILITY:
General Inclusion Criteria

* Age >= 18 years
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Fellow eye (if not a study eye) meets criteria.
* Able and willing to provide informed consent. Study Eye Inclusion Criteria Subjects may have one or two study eyes. Subjects with two study eyes will be randomly assigned to receive sham injection at baseline and 4 weeks in one eye and either ranibizumab or triamcinolone in the other eye.
* Presence of severe nonproliferative or proliferative diabetic retinopathy for which investigator intends to complete panretinal photocoagulation within 49 days after randomization.
* Diabetic macular edema(DME) present on clinical exam and central subfield thickness on Optical Coherence Tomography (OCT) >250 microns, within 8 days of randomization.
* Best corrected Electronic-Early Treatment Diabetic Retinopathy Study visual acuity letter score >=24 (i.e., 20/320 or better), within 8 days of randomization.
* Media clarity, pupillary dilation, and subject cooperation sufficient to administer panretinal photocoagulation and obtain adequate fundus photographs and OCT.
* If prior macular photocoagulation has been performed, the investigator believes that the study eye may possibly benefit from additional focal photocoagulation.

General Exclusion Criteria

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
* Known allergy to any component of the study drugs.
* Blood pressure > 180/110 (systolic above 180 or diastolic above 110).
* Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
* Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Systemic anti-vascular endothelial growth factor(VEGF) or pro-VEGF treatment within 4 months prior to randomization.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 12 months of the study.

Study Eye Exclusion Criteria, Study eye only:

* Prior panretinal photocoagulation that was sufficiently extensive that the investigator does not believe that at least 1200 additional burns are needed or possible within 49 days after randomization.
* Macular edema is considered to be due to a cause other than diabetic macular edema.
* An ocular condition is present such that, in the opinion of the investigator, preventing visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, non-retinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., retinal vein or artery occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of treatment for DME at any time in the past 4 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-VEGF drugs, or any other treatment).
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
* History of Yttrium Aluminum Garnet capsulotomy performed within 2 months prior to randomization.
* Aphakia.
* Intraocular pressure >= 25 mmHg.
* History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion criterion).
* History of steroid-induced intraocular pressure elevation that required intraocular pressure-lowering treatment.
* History of prior herpetic ocular infection.
* Exam evidence of ocular toxoplasmosis.
* Exam evidence of pseudoexfoliation.
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

Fellow Eye Criteria

* Intraocular pressure < 25 mmHg.
* No history of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion criterion).
* No history of steroid-induced intraocular pressure elevation that required intraocular pressure-lowering treatment.
* No exam evidence of pseudoexfoliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J. Brucker, M.D., Study Chair — Scheie Eye Institute; Joseph Googe, Jr., M.D., Study Chair — Southeastern Retina Associates, P.C.
Locations (56):
- United States (56):
  - Sall Research Medical Center, Artesia, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of California, Irvine, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Eldorado Retina Associates, P.C., Louisville, Colorado
  - Retina Vitreous Consultants, Fort Lauderdale, Florida
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Vitreoretinal Consultants, Bangor, Maine
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Ophthalmological Institute at Johns Hopkins, Baltimore, Maryland
  - Retina Consultants of Delmarva, P.A., Salisbury, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Retina Center, PA, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - University of North Carolina, Dept of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Horizon Eye Care, PA, Charlotte, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - OSU Eye Physicians and Surgeons, LLC., Dublin, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Consultants, Providence, Rhode Island
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - West Texas Retina Consultants P.A., Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Virginia Retina Center, Leesburg, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin

REFERENCES:
- [Background] Diabetic Retinopathy Clinical Research Network; Writing Committee; Aiello LP, Beck RW, Bressler NM, Browning DJ, Chalam KV, Davis M, Ferris FL 3rd, Glassman AR, Maturi RK, Stockdale CR, Topping TM. Rationale for the diabetic retinopathy clinical research network treatment protocol for center-involved diabetic macular edema. Ophthalmology. 2011 Dec;118(12):e5-14. doi: 10.1016/j.ophtha.2011.09.058. PMID 22136692
- [Background] Glassman AR, Stockdale CR, Beck RW, Baker C, Bressler NM; Diabetic Retinopathy Clinical Research Network. Evaluation of masking study participants to intravitreal injections in a randomized clinical trial. Arch Ophthalmol. 2012 Feb;130(2):190-4. doi: 10.1001/archophthalmol.2011.387. PMID 22332211
- [Background] Bressler SB, Qin H, Beck RW, Chalam KV, Kim JE, Melia M, Wells JA 3rd; Diabetic Retinopathy Clinical Research Network. Factors associated with changes in visual acuity and central subfield thickness at 1 year after treatment for diabetic macular edema with ranibizumab. Arch Ophthalmol. 2012 Sep;130(9):1153-61. doi: 10.1001/archophthalmol.2012.1107. PMID 22965591
- [Background] Bressler SB, Qin H, Melia M, Bressler NM, Beck RW, Chan CK, Grover S, Miller DG; Diabetic Retinopathy Clinical Research Network. Exploratory analysis of the effect of intravitreal ranibizumab or triamcinolone on worsening of diabetic retinopathy in a randomized clinical trial. JAMA Ophthalmol. 2013 Aug;131(8):1033-40. doi: 10.1001/jamaophthalmol.2013.4154. PMID 23807371
- [Background] Bressler SB, Almukhtar T, Aiello LP, Bressler NM, Ferris FL 3rd, Glassman AR, Greven CM; Diabetic Retinopathy Clinical Research Network. Green or yellow laser treatment for diabetic macular edema: exploratory assessment within the Diabetic Retinopathy Clinical Research Network. Retina. 2013 Nov-Dec;33(10):2080-8. doi: 10.1097/IAE.0b013e318295f744. PMID 23792486
- [Background] Bressler SB, Almukhtar T, Bhorade A, Bressler NM, Glassman AR, Huang SS, Jampol LM, Kim JE, Melia M; Diabetic Retinopathy Clinical Research Network Investigators. Repeated intravitreous ranibizumab injections for diabetic macular edema and the risk of sustained elevation of intraocular pressure or the need for ocular hypotensive treatment. JAMA Ophthalmol. 2015 May;133(5):589-97. doi: 10.1001/jamaophthalmol.2015.186. PMID 25719991
- [Background] Bressler SB, Melia M, Glassman AR, Almukhtar T, Jampol LM, Shami M, Berger BB, Bressler NM; Diabetic Retinopathy Clinical Research Network. RANIBIZUMAB PLUS PROMPT OR DEFERRED LASER FOR DIABETIC MACULAR EDEMA IN EYES WITH VITRECTOMY BEFORE ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR THERAPY. Retina. 2015 Dec;35(12):2516-28. doi: 10.1097/IAE.0000000000000617. PMID 26035510
- [Result] Elman MJ, Bressler NM, Qin H, Beck RW, Ferris FL 3rd, Friedman SM, Glassman AR, Scott IU, Stockdale CR, Sun JK; Diabetic Retinopathy Clinical Research Network. Expanded 2-year follow-up of ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):609-14. doi: 10.1016/j.ophtha.2010.12.033. PMID 21459214
- [Result] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Result] Diabetic Retinopathy Clinical Research Network; Elman MJ, Qin H, Aiello LP, Beck RW, Bressler NM, Ferris FL 3rd, Glassman AR, Maturi RK, Melia M. Intravitreal ranibizumab for diabetic macular edema with prompt versus deferred laser treatment: three-year randomized trial results. Ophthalmology. 2012 Nov;119(11):2312-8. doi: 10.1016/j.ophtha.2012.08.022. Epub 2012 Sep 19. PMID 22999634
- [Result] Bressler SB, Glassman AR, Almukhtar T, Bressler NM, Ferris FL, Googe JM Jr, Gupta SK, Jampol LM, Melia M, Wells JA 3rd; Diabetic Retinopathy Clinical Research Network. Five-Year Outcomes of Ranibizumab With Prompt or Deferred Laser Versus Laser or Triamcinolone Plus Deferred Ranibizumab for Diabetic Macular Edema. Am J Ophthalmol. 2016 Apr;164:57-68. doi: 10.1016/j.ajo.2015.12.025. Epub 2016 Jan 21. PMID 26802783
- [Result] Elman MJ, Ayala A, Bressler NM, Browning D, Flaxel CJ, Glassman AR, Jampol LM, Stone TW; Diabetic Retinopathy Clinical Research Network. Intravitreal Ranibizumab for diabetic macular edema with prompt versus deferred laser treatment: 5-year randomized trial results. Ophthalmology. 2015 Feb;122(2):375-81. doi: 10.1016/j.ophtha.2014.08.047. Epub 2014 Oct 28. PMID 25439614
- [Derived] Gangaputra S, Almukhtar T, Glassman AR, Aiello LP, Bressler N, Bressler SB, Danis RP, Davis MD; Diabetic Retinopathy Clinical Research Network. Comparison of film and digital fundus photographs in eyes of individuals with diabetes mellitus. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6168-73. doi: 10.1167/iovs.11-7321. PMID 21571677
- [Derived] Bhavsar AR, Googe JM Jr, Stockdale CR, Bressler NM, Brucker AJ, Elman MJ, Glassman AR; Diabetic Retinopathy Clinical Research Network. Risk of endophthalmitis after intravitreal drug injection when topical antibiotics are not required: the diabetic retinopathy clinical research network laser-ranibizumab-triamcinolone clinical trials. Arch Ophthalmol. 2009 Dec;127(12):1581-3. doi: 10.1001/archophthalmol.2009.304. PMID 20008710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from 1 clinical site where a majority of eyes were judged not to meet the Optical Coherence Tomography eligibility criterion of central subfield >=250 microns when graded manually at a central reading center (14 eyes of 10 subjects) are excluded from all analysis except for safety data.
Pre-assignment Details: Participants with 2 study eyes enrolled each eye in a different arm. Each treatment arm includes no more than 1 study eye for a given participant, and thus the numbers of eyes is equal to the number of participants in each arm.
Groups:
- 0.5mg Ranibizumab: Intravitreal injections of 0.5mg Ranibizumab at baseline and at 4 weeks
- 4-mg Triamcinolone Acetonided: 4-mg Triamcinolone Acetonide at baseline and sham injection at 4 weeks
Period: Overall Study
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Started | 123 | 113 | 109
Completed | 118 | 103 | 105
Not Completed | 5 | 10 | 4
Not completed — Death | 1 | 2 | 1
Not completed — Missed Visit | 3 | 5 | 1
Not completed — Dropped | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided | Total
Number analyzed (Participants) | 123 | 113 | 109 | 345
Age, Customized [Median (Inter-Quartile Range); unit: years] | 54 [45 to 61] | 57 [48 to 64] | 58 [49 to 64] | 56 [45 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 44 | 136
  Male | 79 | 65 | 65 | 209
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 11 | 15 | 18 | 44
  White | 76 | 72 | 61 | 209
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
  Hispanic or Latino | 31 | 23 | 27 | 81
Optical coherence tomography subretinal fluid present (questionable or definite) [Number; unit: Eyes] — Based on standard reading center grading
  Eyes
    Yes | 30 | 31 | 32 | 93
    No | 93 | 82 | 77 | 252
Classification of diabetic macular edema on clinical exam [Number; unit: Eyes]
  Predominantly Focal' | 37 | 19 | 27 | 83
  Neither perdominantly focal or diffuse | 18 | 25 | 14 | 57
  Predominantly diffuse | 68 | 69 | 68 | 205
Intraocular Pressure [Median (Inter-Quartile Range); unit: mmHg] | 15 [13 to 18] | 16 [14 to 18] | 15 [13 to 18] | 15 [13 to 18]
Diabetes Type [Number; unit: Participants]
  Type 1 | 20 | 13 | 12 | 45
  Type 2 | 101 | 93 | 95 | 289
  Uncertain | 2 | 7 | 2 | 11
Duration of diabetes [Median (Inter-Quartile Range); unit: Years] | 15 [8 to 21] | 15 [10 to 21] | 15 [10 to 19] | 15 [8 to 21]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Percentage] — Missing hemoglobin A1c data for study participants in the sham, ranibizumab, and triamcinolone, respectively: 4, 10, 7
  Percentage | 7.9 [7.0 to 9.6] | 8.1 [7.1 to 9.9] | 8.1 [7.0 to 9.7] | 8.0 [7.0 to 9.9]
Prior Cardiovascular event [Number; unit: Participants]
  Yes | 21 | 35 | 28 | 84
  No | 102 | 78 | 81 | 261
Hypertension [Number; unit: Participants]
  Yes | 97 | 88 | 82 | 267
  No | 26 | 25 | 27 | 78
Number of study eyes [Number; unit: Participants]
  1 study eye | 97 | 100 | 96 | 293
  2 study eyes | 26 | 13 | 13 | 52
Prior Panretinal scatter photocoagulation [Number; unit: Eyes]
  Yes | 16 | 20 | 19 | 55
  No | 107 | 93 | 90 | 290
prior treatment for diabetic macular edema [Number; unit: Eyes]
  Yes | 80 | 75 | 72 | 227
  No | 43 | 38 | 37 | 118
Prior laser for diabetic macular edema [Number; unit: Eyes]
  Yes | 40 | 33 | 36 | 109
  No | 83 | 80 | 73 | 236
Prior intravitreal triamcinolone for diabetic macular edema [Number; unit: Eyes]
  Yes | 1 | 9 | 3 | 13
  No | 122 | 104 | 106 | 332
Prior vitrectomy for diabetic macular edema [Number; unit: Eyes]
  Yes | 2 | 0 | 0 | 2
  No | 121 | 113 | 109 | 343
Prior peribulbar triamcinolone for diabetic macular edema [Number; unit: Eyes]
  Yes | 1 | 0 | 1 | 2
  No | 122 | 113 | 108 | 343
prior anti- vascular endothelial growth factor for diabetic macular edema [Number; unit: Eyes]
  Yes | 6 | 1 | 3 | 10
  No | 117 | 112 | 106 | 335
Currently on intraocular pressure lowering medication for glaucoma or ocular hypertension [Number; unit: Eyes]
  Yes | 0 | 3 | 0 | 3
  No | 123 | 110 | 109 | 342
Lens status (clinical examination) [Number; unit: Eyes]
  Phakic | 111 | 91 | 99 | 301
  Pseudophakic | 12 | 22 | 10 | 44
Baseline visual acuity by randomization strata [Median (Inter-Quartile Range); unit: Letter Score] — Visual Acuity was measured with the Electronic Early Treatment Study (E-ETDRS) visual acuity test. Unit of measure is based on the E-ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
  Letter Score | 67 [52 to 75] | 68 [56 to 75] | 67 [59 to 75] | 67 [52 to 75]
Central subfield thickness on optical coherence tomography [Median (Inter-Quartile Range); unit: Microns] | 355 [285 to 510] | 352 [283 to 476] | 359 [271 to 472] | 355 [283 to 510]
Retinal volume on optical coherence tomography [Median (Inter-Quartile Range); unit: cubic millimetre] | 9.4 [8.4 to 10.6] | 9.2 [8.3 to 11.0] | 9.1 [8.1 to 10.0] | 9.2 [8.1 to 11]
Optical coherence tomography cystoid abnormality (questionable or definite) [Number; unit: Eyes] — From reading center grading.
  Eyes
    Yes | 108 | 96 | 96 | 300
    No | 15 | 17 | 13 | 45
Early Treatment Diabetic Retinopath Study Retinopathy severity level from photograph grading [Number; unit: Eyes] — Criteria are based on the ETDRS fundus photographic risk factors for the progression of diabetic retinopathy. ETDRS report no. 12. Ophthalmology 1991; 98:823-833
  Eyes
    Level 35, 43 (Mild/Moderate NPDR) | 6 | 5 | 6 | 17
    Level 47 (Moderately severe NPDR) | 26 | 15 | 10 | 51
    Level 53 (Severe NPDR) | 5 | 6 | 5 | 16
    Level 60 (Prior PRP without active neovascularizat | 2 | 4 | 3 | 9
    Level 61 (Mild/Moderate PDR) | 48 | 36 | 38 | 122
    Level 71, 75 (High-risk PDR) | 32 | 43 | 43 | 118
    cannot grade | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Electronic Early Treatment Diabetic Retinopathy Study Visual Acuity Letter Score From Baseline to 14 Weeks
Description: Visual Acuity was measured with the Electronic Early Treatment Study (E-ETDRS) visual acuity test. Unit of measure is based on the E-ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
Time Frame: baseline to 14 weeks
Population: Participants with 2 study eyes enrolled each eye in a different arm. Each arm includes no more than 1 study eye for a given participant, and thus the numbers of eyes is equal to the number of participants in each arm. Analysis followed intention to treat principle; eyes without 14-week data, the Last Observation Carried Forward method was used.
Measure: Mean (Standard Deviation); unit: Letter Score
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 123 | 113 | 109
Letter Score | -4 (14) | 1 (11) | 2 (11)
Statistical Analysis 1: Comparison: Sham Injection vs 0.5mg Ranibizumab; Test type: Superiority or Other; p < .001, ANCOVA — adjusted for baseline visual acuity, number of planned panretinal photocoagulation sittings, and correlation between two study eyes; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [2.2 to 9.0] — adjusted for multiple comparison
Statistical Analysis 2: Comparison: Sham Injection vs 4-mg Triamcinolone Acetonided; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.7, 95% CI 2-sided [3.2 to 10.1] — adjusted for multiple comparisons

2. Secondary Outcome: Additional Treatments for Diabetic Macular Edema
Description: Each combination of treatment is only counted once per treatment eye. Participants could have 2 study eyes, with random assignments to different treatments.
Time Frame: 14 weeks to 56-weeks
Measure: Number; unit: Eyes
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 123 | 113 | 109
Eyes
  Bevacizumab | 14 | 12 | 9
  Ranibizumab | 1 | 0 | 3
  Triamcinolone | 3 | 8 | 2
  Pegaptanib | 0 | 0 | 3
  Laser | 31 | 10 | 21
  Vitrectomy | 2 | 1 | 0
  Bevacizumab plus Triamcinolone | 2 | 0 | 2
  Ranibizumab plus Triamcinolone | 0 | 1 | 0
  Bevacizumab plus laser | 8 | 5 | 0
  Ranibizumab plus laser | 0 | 3 | 0
  Triamcinolone plus laser | 7 | 4 | 5
  Pegaptanib plus laser | 1 | 0 | 0
  Triamcinolone plus vitrectomy | 0 | 1 | 0
  Pegaptanib plus vitrectomy | 0 | 1 | 0
  Triamcinolone plus laser plus vitrectomy | 0 | 1 | 0
  Bevacizumab plus triamcinolone plus laser | 2 | 1 | 0

3. Secondary Outcome: Change in Optical Coherence Tomography Central Subfield Thickness
Time Frame: Baseline to 14 weeks
Population: Participants with two study eyes enrolled each eye in a different treatment group. Therefore, each treatment group/arm includes no more than one study eye for a given participant, and thus the numbers of eyes is equal to the number of participants in each arm.
Measure: Median (Inter-Quartile Range); unit: Microns
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 123 | 113 | 109
Microns | 362 [287 to 484] | 312 [259 to 453] | 265 [230 to 304]
Statistical Analysis 1: Comparison: Sham Injection vs 0.5mg Ranibizumab; Test type: Superiority or Other; p < .01, ANCOVA — Adjusted for baseline optical coherence tomography retinal thickness and visual acuity, number of planned panretinal photocoagulation sittings, and correlation between 2 study eyes; Mean Difference (Final Values) = -35, 95% CI 2-sided [-64 to -6] — adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Sham Injection vs 4-mg Triamcinolone Acetonided; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -100, 95% CI 2-sided [-128 to -71] — adjusted for multiple comparisons

4. Secondary Outcome: Total Optical Coherence Tomography Retinal Volume
Description: Missing/ungradable as follows: Sham = 49, Ranibizumab = 37, Triamcinolone = 39. Visits occured between 70 days and 153 days from randomization adjusted for baseline optical coherence tomography (OCT) retinal volume, OCT retinal thickness and visual acuity, number of planned panretinal photocoagulation sittings, and correlation between 2 study eyes. Confidence intervals are adjusted for multiple comparisons.
Time Frame: Baseline to 14-weeks
Population: Participants with 2 study eyes enrolled each eye in a different arm. Therefore, each arm includes no more than 1 eye for a given participant, and thus the numbers of eyes is equal to number of participants.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 69 | 66 | 66
mm^3 | 9.7 (1.8) | 9.3 (1.9) | 7.9 (1.0)

5. Secondary Outcome: Change in Visual Acuity From Baseline
Description: as for outcome 1
Time Frame: baseline to 56-weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Letter Score
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 111 | 95 | 93
Letter Score | -6 (17) | -4 (21) | -5 (16)
Statistical Analysis 1: Comparison: Sham Injection vs 0.5mg Ranibizumab; Test type: Superiority or Other; p = 0.44, ANCOVA — Adjusted for baseline visual acuity, number of planned panretinal photocoagulation sittings, and correlation between 2 study eyes; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-3.7 to 7.5] — adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Sham Injection vs 4-mg Triamcinolone Acetonided; Test type: Superiority or Other; p = 0.63, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-4.4 to 6.8] — adjusted for multiple comparisons

6. Secondary Outcome: Eyes With Anti-vascular Endothelial Growth Factor Treatment for Diabetic Macular Edema
Time Frame: 14 weeks to 56-weeks
Population: as for outcome 3
Measure: Number; unit: Eyes
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 123 | 113 | 109
Eyes | 28 | 23 | 17

7. Secondary Outcome: Number of Eyes With Additional Number of Treatments for Diabetic Macular Edema
Description: Treatments include any type or combination of treatment for diabetic macular edema. Eyes were only counted once, when receiving a combination of treatments.
Time Frame: 14 weeks to 56-weeks
Population: as for outcome 3
Measure: Number; unit: Eyes
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 123 | 113 | 109
Eyes | 71 | 48 | 45

8. Secondary Outcome: Change in Optical Coherence Tomography Retinal Volume
Description: Missing or un-gradable data as follows for the sham plus focal/grid/panretinal photocoagulation laser, triamcinolone plus focal/grid panretinal photocoagulation laser, and Ranibizumab groups were 49, 37, and 39, respectively
Time Frame: Baseline to 14 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Number analyzed (Participants) | 69 | 66 | 66
mm^3 | 0.1 (1.1) | -0.4 (1.3) | -1.3 (1.3)
Statistical Analysis 1: Comparison: Sham Injection; Test type: Superiority or Other; p = 0.001, ANCOVA — adjusted for baseline retinal volume, optical coherence tomography retinal thickness and visual acuity, number of planned panretinal photocoagulation sittings, and correlation between 2 study eyes; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.2] — adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Sham Injection vs 4-mg Triamcinolone Acetonided; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.1 to -1.3] — adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Through 14-week Primary outcome visit
Description: Data from 1 clinical site where a majority of eyes were judged not to meet the Optical Coherence Tomography eligibility criterion of central subfield >=250 microns when graded manually at a central reading center (14 eyes of 10 subjects) are excluded from all analysis except for safety data.
Arm/Group | Sham Injection | 0.5mg Ranibizumab | 4-mg Triamcinolone Acetonided
Serious Adverse Events (participants affected / at risk) | 11/133 | 15/116 | 12/115
Other Adverse Events (participants affected / at risk) | 57/133 | 50/116 | 66/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=133) | 0.5mg Ranibizumab (N=116) | 4-mg Triamcinolone Acetonided (N=115)
Abdominal pain (General disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cellulitis (General disorders) | 0 | 1 | 0
Cerebrovascular accident (General disorders) | 1 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0
Cholelithiasis (Gastrointestinal disorders) | 0 | 0 | 1
Convulsion (General disorders) | 0 | 0 | 1
Coronary arterial stant insertion (Surgical and medical procedures) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Death (General disorders) | 1 | 1 | 1
Diabetes mellitus (General disorders) | 1 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Endophthalmitis (Eye disorders) | 0 | 1 | 0
Heart rate decreased (Cardiac disorders) | 0 | 1 | 0
Hypertension (General disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Ischaemic stroke (General disorders) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Nausea (General disorders) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Renal failure (Endocrine disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Transient ischaemic attach (Cardiac disorders) | 1 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Vomiting (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=133) | 0.5mg Ranibizumab (N=116) | 4-mg Triamcinolone Acetonided (N=115)
Conjunctival haemorrhage (Eye disorders) | 2 | 11 | 8
Eye pain (Eye disorders) | 11 | 7 | 6
headache (General disorders) | 7 | 7 | 5
Intraocular pressure increase (Eye disorders) | 1 | 0 | 11
Myodesopsia (Eye disorders) | 5 | 7 | 10
Vision Blurred (Eye disorders) | 13 | 8 | 9
Vitreous floaters (Eye disorders) | 3 | 4 | 10
Vitreous haemorrhage (Eye disorders) | 15 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less